CLINICAL TRIAL: NCT02952742
Title: Black Cohosh (Actaea Racemosa) for Hot Flashes in Prostate Cancer Patients on Androgen Deprivation Therapy: A Randomized, Placebo-Controlled, Double-Blind Clinical Trial
Brief Title: Black Cohosh for Host Flashes Due to Androgen Deprivation Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding support
Sponsor: Midwestern Regional Medical Center (Other)
Responsible Party: Principal Investigator, Evan Pisick, Medical Oncologist, Midwestern Regional Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MZ2016003
Record Dates: First submitted 2016-03-15; First posted 2016-11-02 (Estimated); Last update posted 2017-12-26 (Actual); Status verified 2017-12

CONDITIONS: Hot Flashes
MeSH Terms: conditions — Hot Flashes | interventions — black cohosh root extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Black Cohosh Therapy (Experimental): Black Cohosh will be provided in 250mg capsules. Subjects will take 2 capsules by mouth daily for a total daily dose of 500 mg. Subject's will remain on this study arm for 8 weeks.
  Interventions: Drug: Black Cohosh
- Placebo (Placebo Comparator): Subjects will take 2 capsules, identical to the Black Cohosh capsules, by mouth each. Subject's will remain on this study arm for 8 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Black Cohosh — Vital Nutrients Black Cohosh Extract
  Other Names: Actaea racemosa
  Arms: Black Cohosh Therapy
Other: Placebo — Inactive comparator resembling the Black Cohosh formulation in appearance. Ingredients include: cellulose; caramel color; powdered yellow dye; and powdered red dye.
  Arms: Placebo

SUMMARY:
This is a randomized, placebo-controlled crossover study. Participants will be actively participating in the study for 6 months, and enrolled in the study for up to 1 year. During the first phase of the study, the participants will be randomized into either the placebo group or treatment group for 8 weeks following 1 week of baseline data collection (no treatment). Following this first phase, a no-treatment washout period of at least 3 weeks will be implemented for all participants. After the washout period, the randomized groups will switch from treatment to placebo group, or placebo to treatment group for an additional 8 week period. Hot flash frequency and severity will be documented using a daily hot flash diary and calculated using the Hot Flash Score questionnaire. The impact on quality of life will be documented by weekly Hot Flash Related Daily Interference Scale (HFRDIS) questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand English or be wiling to use a trained interpreter
* Diagnosis of prostate cancer
* Receiving either Leuprolide or Degarelix,for prostate cancer treatment
* Currently experiencing a minimum of 3 self-reported hot flashes within a 24 hour period
* Eastern Cooperative Oncology Group (ECOG) performance status score < 2
* Life expectancy >3 months.
* No grade 3 or higher toxicity from prior cancer therapies unless judged by the principal investigator to be clinically irrelevant to study procedures
* At least four (4) weeks following prior major surgery
* Serum testosterone concentration below castrate level (< 30 ng/dL) at time of recruitment
* Willing to provide written informed consent for participation in the study

Exclusion Criteria:

* Concurrent severe illness effecting ECOG performance status or life expectancy as determined by the principal investigator
* Hormone refractory patients. Patients taking Enzalutamide or Abiraterone.
* Active infection
* Psychiatric illness or social situation that would limit safety and compliance with study requirements
* Currently taking any pharmaceutical medications that have potential interactions with black cohosh as determined by the principal investigator
* Currently taking any supplements that have potential interactions with black cohosh as determined by the principal investigator
* Currently receiving any treatment for hot flashes or planning to initiate any treatment for hot flashes other than with study supplementation
* ALT, AST, or Bilirubin > 2 times their normal laboratory values in the past 3 months
* Inability to complete the informed consent process or adhere to the protocol treatment plan.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2018-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Frequency of hot flashes as calculated from self reported questionnaire | Daily assessments throughout the study (assessed for up to 16 weeks)
  Subjects will record the number and timing of their on the Hot Flash Related Daily Interference (HFRDIS) questionnaire each week during the study.

SECONDARY OUTCOMES:
Severity of hot flashes as calculated from self reported questionnaire | Daily assessments throughout the study (assessed for up to 16 weeks)
  Subjects will record the intensity of their hot flashes on the Hot Flash Related Daily Interference (HFRDIS) questionnaire each day during the study.
Quality of life as recorded from self reported questionnaire | Daily assessments throughout the study (assessed for for up to 16 weeks)
  Subjects will answer questions regarding the impact of their hot flashes on the Hot Flash Related Daily Interference (HFRDIS) questionnaire each day during the study.
Measurement of serum testosterone | From the beginning of treatment to the end of the 8-week treatment phase (up to 16 weeks due to cross-over of study arms)
  The effect of Black Cohosh on serum testosterone will be measured at the end of each 8-week treatment cycle.
Measurement of serum aspartate aminotransferase (AST) | From the beginning of treatment to the end of the 8-week treatment phase (up to 16 weeks due to cross-over of study arms)
  The effect of Black Cohosh on AST will be measured at the end of each 8-week treatment cycle.
Measurement of serum alanine aminotransferase (ALT) | From the beginning of treatment to the end of the 8-week treatment phase (up to 16 weeks due to cross-over of study arms)
  The effect of Black Cohosh on serum ALT will be measured at the end of each 8-week treatment cycle.
Measurement of serum bilirubin | From the beginning of treatment to the end of the 8-week treatment phase (up to 16 weeks due to cross-over of study arms)
  The effect of Black Cohosh on serum bilirubin will be measured at the end of each 8-week treatment cycle.
Measurement of serum Prostate Specific Antigen (PSA) | From the beginning of treatment to the end of the 8-week treatment phase (up to 16 weeks due to cross-over of study arms)
  The effect of Black Cohosh on serum PSA will be measured at the end of each 8-week treatment cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Evan Pisick, MD, Principal Investigator — Midwestern Regional Medical Center

IPD SHARING:
Plan to Share IPD: Undecided